CLINICAL TRIAL: NCT00127166
Title: A Multicenter, Double-Blind, Randomized, Crossover Design Study to Evaluate the Effect of Montelukast Vs. Salmeterol on the Inhibition of Exercise-Induced Bronchoconstriction in Asthmatic Patients Aged 6-14 Years
Brief Title: Two Investigational Drugs in the Prevention of Airway Constriction Brought on by Exercise in Participants With Asthma (0476-911)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-911; 2004_006 (Other: Merck Registration Number)
Record Dates: First submitted 2005-06-30; First posted 2005-08-05 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Exercise Induced Asthma
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — montelukast; Salmeterol Xinafoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast/Salmeterol (Experimental): Period I - Montelukast 5 milligrams (mg) oral tablet once daily and Salmeterol matching placebo dry powder inhaler (DPI) twice daily for 4 weeks followed by a 2-week washout period (salmeterol matching placebo + montelukast matching placebo). Period II - Montelukast matching placebo oral tablet once daily and Salmeterol DPI 50 micrograms (mcg) twice daily for 4 weeks. Inhaled Fluticasone 100 mcg twice daily throughout the study.
  Interventions: Drug: Montelukast sodium; Drug: Salmeterol xinafoate; Drug: Fluticasone propionate; Drug: Montelukast matching placebo; Drug: Salmeterol matching placebo
- Salmeterol/Montelukast (Experimental): Period I - Montelukast matching placebo oral tablet once daily and Salmeterol DPI 50 mcg twice daily for 4 weeks followed by a 2-week washout period (salmeterol matching placebo + montelukast matching placebo). Period II - Montelukast 5 mg oral tablet once daily and Salmeterol matching placebo DPI twice daily for 4 weeks. Inhaled Fluticasone 100 mcg twice daily throughout the study.
  Interventions: Drug: Montelukast sodium; Drug: Salmeterol xinafoate; Drug: Fluticasone propionate; Drug: Montelukast matching placebo; Drug: Salmeterol matching placebo

INTERVENTIONS:
Drug: Montelukast sodium — Montelukast 5 mg chewable tablet once daily
Drug: Salmeterol xinafoate — Salmeterol 50 mcg dry powder per actuation inhaled twice daily
Drug: Fluticasone propionate — Fluticasone (50 mcg per actuation) 100 mcg inhaled twice daily
Drug: Montelukast matching placebo — Matching placebo to montelukast oral tablet administered once daily.
Drug: Salmeterol matching placebo — Matching placebo to salmeterol dry powder for inhalation administered twice daily

SUMMARY:
The purpose of this study is to determine the effect of four weeks of treatment with two investigational drugs (oral versus inhaled administration) plus an inhaled medication in the treatment of airway constriction brought on by exercise in participants with asthma.

ELIGIBILITY:
Inclusion Criteria:

* 6-14 year old children with a history of asthma for at least 12 months
* must demonstrate airway constriction brought on by exercise

Exclusion Criteria:

* is taking any medications that are not allowed in the study

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2005-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fogel RB, Rosario N, Aristizabal G, Loeys T, Noonan G, Gaile S, Smugar SS, Polos PG. Effect of montelukast or salmeterol added to inhaled fluticasone on exercise-induced bronchoconstriction in children. Ann Allergy Asthma Immunol. 2010 Jun;104(6):511-7. doi: 10.1016/j.anai.2009.12.011. PMID 20568384

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter Study (30 Ex-US sites) Study Initiation Date: December 22, 2005 Study Completion Date: November 14, 2008
Pre-assignment Details: For randomization, patients fulfilled the following criteria:
  1. Forced Expiratory Volume in one second (FEV1) ≥70% predicted while withholding beta (β)-agonist for at least 6 hours
  2. Exercise-induced bronchoconstriction (EIB) showing FEV1 ≥15% reduction from baseline while on inhaled corticosteroids demonstrated twice during the run-in period.
Groups:
- Montelukast / Salmeterol: Period I- Montelukast 5 milligrams (mg) oral tablet once daily and Salmeterol matching placebo dry powder inhaler (DPI) twice daily for 4 weeks followed by a 2-week washout period (salmeterol matching placebo + montelukast matching placebo). Period II- Montelukast matching placebo oral tablet once daily and Salmeterol DPI 50 micrograms (mcg) twice daily for 4 weeks. Inhaled Fluticasone 100 mcg twice daily throughout the study.
- Salmeterol / Montelukast: Period I- Montelukast matching placebo oral tablet once daily and Salmeterol DPI 50 mcg twice daily for 4 weeks followed by a 2-week washout period (salmeterol matching placebo + montelukast matching placebo). Period II- Montelukast 5 mg oral tablet once daily and Salmeterol matching placebo DPI twice daily for 4 weeks. Inhaled Fluticasone 100 mcg twice daily throughout the study.
Period: Period I
Arm/Group | Montelukast / Salmeterol | Salmeterol / Montelukast
Started | 78 | 76
Completed | 75 | 74
Not Completed | 3 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Patient did not meet inclusion criteria | 1 | 0
Period: Washout Period
Arm/Group | Montelukast / Salmeterol | Salmeterol / Montelukast
Started | 75 | 74
Completed | 75 | 73
Not Completed | 0 | 1
Not completed — Patient did not meet inclusion criteria | 0 | 1
Period: Period II
Arm/Group | Montelukast / Salmeterol | Salmeterol / Montelukast
Started | 75 | 73
Completed | 72 | 73
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Patient did not perform Visit 6 exercise | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast / Salmeterol | Salmeterol / Montelukast | Total
Number analyzed (Participants) | 78 | 76 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (2.0) | 9.8 (2.0) | 10.0 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 30 | 65
  Male | 43 | 46 | 89
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black | 11 | 7 | 18
  White | 38 | 41 | 79
  Other | 28 | 28 | 56
Area Under the Curve from 0 to 20 minutes (AUC0-20) [Mean (Standard Deviation); unit: Percent times Minutes] — Area Under the Curve for percent-change from pre-exercise baseline FEV1 in liters, from 0 to 20 minutes (AUC0-20)
  Percent times Minutes | 320.08 (208.62) | 317.74 (165.71) | 318.93 (188.06)
Avg %-change from pre-exercise baseline FEV1 after 1st β-agonist use & prior to 2nd β-agonist use [Mean (Standard Deviation); unit: Percent change from baseline] | 1.36 (10.99) | 4.78 (10.92) | 3.05 (11.05)
Maximum FEV1 percent predicted [Mean (Standard Deviation); unit: Percent of predicted value] | 99.88 (32.45) | 100.54 (15.61) | 100.21 (25.49)
Maximum percent fall in FEV1 after exercise [Mean (Standard Deviation); unit: Percent change from baseline] | 24.77 (10.25) | 25.42 (9.04) | 25.09 (9.65)
Time to recovery [Mean (Standard Deviation); unit: Minutes] — Montelukast / Salmeterol, n=71; Salmeterol / Montelukast, n=70
  Minutes | 23.53 (10.53) | 21.51 (8.30) | 22.53 (9.51)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Post-exercise Percent (%) Fall in FEV1
Description: The effect of four weeks of treatment with oral montelukast plus inhaled fluticasone, and inhaled salmeterol plus inhaled fluticasone on EIB as measured by the maximum post-exercise percent fall (relative to pre-exercise baseline) in FEV1.
Time Frame: 4 weeks (Weeks 0 to 4 or Weeks 6 to 10)
Population: The primary efficacy analysis was based on the full analysis set (FAS) population which included all randomized participants who took at least one dose of post randomization study drug and had a measurement for analysis available in both treatment periods of the cross-over design.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Groups:
- Montelukast: Montelukast 5 mg oral tablet once daily, inhaled Fluticasone 100 mcg twice daily.
- Salmeterol: Salmeterol DPI 50 mcg twice daily, inhaled Fluticasone 100 mcg twice daily.
Arm/Group | Montelukast | Salmeterol
Number analyzed (Participants) | 144 | 144
Percent change from baseline | 10.57 [8.86 to 12.27] | 13.82 [12.11 to 15.52]
Statistical Analysis 1: Comparison: Montelukast vs Salmeterol; Test type: Superiority or Other; p = 0.009, ANOVA; Model terms: participant, treatment and period. The treatment test is adjusted for period; Least squares mean difference = -3.25, 95% CI [-5.66 to -0.84]

2. Secondary Outcome: Area Under the Curve for %-Change From Pre-exercise Baseline FEV1 in Liters (L), From 0 to 20 Minutes (AUC(0-20))
Description: The effect of a four-week treatment course of oral montelukast plus inhaled fluticasone, compared to inhaled salmeterol plus inhaled fluticasone, on the extent and severity of EIB as measured by the area under the curve from 0 to 20 minutes (AUC0-20) for FEV1 percent change from pre-exercise baseline.
Time Frame: 4 weeks (Weeks 0 to 4 or Weeks 6 to 10)
Population: The secondary efficacy analysis was based on the FAS population which included all randomized participants who took at least one dose of post randomization study drug and had a measurement for analysis available in both treatment periods of the cross-over design.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent times Minutes
Arm/Group | Montelukast | Salmeterol
Number analyzed (Participants) | 144 | 144
Percent times Minutes | 116.04 [89.95 to 142.24] | 168.75 [142.56 to 194.95]
Statistical Analysis 1: Comparison: Montelukast vs Salmeterol; Test type: Superiority or Other; p = 0.006, ANOVA; Model terms: participant, treatment and period. The treatment test is adjusted for period; Least squares mean difference = -52.71, 95% CI [-89.76 to -15.66]

3. Secondary Outcome: Maximum FEV1 % Predicted Following First Beta-agonist Use
Description: The effect of a four-week treatment course of oral montelukast plus inhaled fluticasone, compared to inhaled salmeterol plus inhaled fluticasone, on short-acting β-agonist bronchodilation as measured by the maximum FEV1 percent predicted following first β-agonist use.
Time Frame: 4 weeks (Weeks 0 to 4 or Weeks 6 to 10)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of predicted value
Arm/Group | Montelukast | Salmeterol
Number analyzed (Participants) | 144 | 144
Percent of predicted value | 104.03 [102.83 to 105.23] | 99.92 [98.72 to 101.12]
Statistical Analysis 1: Comparison: Montelukast vs Salmeterol; Test type: Superiority or Other; p < 0.001, ANCOVA; Participant, treatment, period & covariate for FEV1 %-predicted Treatment test is adjusted for period & FEV1 %-predicted at pre-exercise baseline; Least squares mean difference = 4.11, 95% CI [2.58 to 5.64]

4. Secondary Outcome: Time to Recovery to Within 5% of Baseline FEV1
Description: The effect of a four-week treatment course of oral montelukast plus inhaled fluticasone, compared to inhaled salmeterol plus inhaled fluticasone, on the extent and severity of EIB as measured by the time to recovery (to within 5 percent of the pre-exercise baseline FEV1) following a standardized exercise challenge.
Time Frame: 4 weeks (Weeks 0 to 4 or Weeks 6 to 10)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Montelukast | Salmeterol
Number analyzed (Participants) | 144 | 144
minutes | 5.9 [0.0 to 19.12] | 11.1 [0.065 to 22.94]
Statistical Analysis 1: Comparison: Montelukast vs Salmeterol; Test type: Superiority or Other; p = 0.035, Cox Proportional Hazards Model; Model terms: treatment and period; Hazard Ratio (HR) = 1.26, 95% CI [1.02 to 1.55] — Dispersion not applicable to time to event data

5. Secondary Outcome: Average (Avg) %-Change in FEV1 After First Beta (β)-Agonist Use and Prior to Second β-agonist Use
Description: The effect of a four-week treatment course of oral montelukast plus inhaled fluticasone, compared to inhaled salmeterol plus inhaled fluticasone, on the extent and severity of EIB as measured by the average percent change in FEV1 after first β-agonist intake and prior to second β-agonist use.
Time Frame: 4 weeks (Weeks 0 to 4 or Weeks 6 to 10)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | Montelukast | Salmeterol
Number analyzed (Participants) | 144 | 144
Percent change from baseline | 6.51 [5.44 to 7.59] | 2.72 [1.64 to 3.79]
Statistical Analysis 1: Comparison: Montelukast vs Salmeterol; Test type: Superiority or Other; p < 0.001, ANOVA; Model terms: participant, treatment and period. The treatment test is adjusted for period; Least squares mean difference = 3.80, 95% CI [2.28 to 5.32]

ADVERSE EVENTS:
Description: 154 participants (pts) enrolled, but only 150 took at least 1 dose of each treatment (tx). 78 pts were in Montelukast (M)/Salmeterol (S) sequence (seq) and 76 in S/M seq. 4 pts in M/S seq only took 1st tx; so 78 took M & 74 took S. 4 different pts in S/M seq only took 1st tx; so 76 took S & 72 took M. Total of 150 pts took M and 150 took S.
Groups:
- Montelukast: Period I- Montelukast 5 milligrams (mg) oral tablet once daily and Salmeterol matching placebo dry powder inhaler (DPI) twice daily for 4 weeks.
  Period II- Montelukast 5 mg oral tablet once daily and Salmeterol matching placebo DPI twice daily for 4 weeks.
  Inhaled Fluticasone 100 mcg twice daily throughout the study.
- Salmeterol: Period I- Montelukast matching placebo oral tablet once daily and Salmeterol DPI 50 mcg twice daily for 4 weeks.
  Period II- Montelukast matching placebo oral tablet once daily and Salmeterol DPI 50 micrograms (mcg) twice daily for 4 weeks.
  Inhaled Fluticasone 100 mcg twice daily throughout the study.
Arm/Group | Montelukast | Salmeterol
Serious Adverse Events (participants affected / at risk) | 1/150 | 1/150
Other Adverse Events (participants affected / at risk) | 27/150 | 21/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (N=150) | Salmeterol (N=150)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (N=150) | Salmeterol (N=150)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Allergy To Plants (Immune system disorders) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Pertussis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (5) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection Viral (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (3) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 2 (2)
Viral Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Ear Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Menstruation Delayed (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.